CLINICAL TRIAL: NCT04665700
Title: Safety, Tolerability and Pharmacokinetics of Single and Multiple Rising Doses of BI 764198 in Japanese Healthy Male Subjects (Double-blind, Randomised, Placebo-controlled Within Dose Groups, Parallel Group Design)
Brief Title: A Study in Healthy Japanese Men to Test How Well Different Doses of BI 764198 Are Tolerated
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1434-0003
Record Dates: First submitted 2020-12-07; First posted 2020-12-14 (Actual); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: Healthy

STUDY DESIGN:
Intervention Model Description: This trial consists of a single dose part and a multiple rising dose (MRD) part. The first dose group is conducted in the single dose part and the second dose group onwards are conducted in the MRD part.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- BI 764198 Single dose part (Experimental)
  Interventions: Drug: BI 764198
- BI 764198 Multiple dose low (Experimental)
  Interventions: Drug: BI 764198
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- BI 764198 Multiple dose medium (Experimental)
  Interventions: Drug: BI 764198
- BI 764198 Multiple dose high (Experimental)
  Interventions: Drug: BI 764198

INTERVENTIONS:
Drug: BI 764198 — BI 764198
  Arms: BI 764198 Multiple dose high; BI 764198 Multiple dose low; BI 764198 Multiple dose medium; BI 764198 Single dose part
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The main objectives of this trial are to investigate safety and tolerability of BI 764198 in healthy male subjects following oral administration of single dose and multiple rising doses per day over 14 days.

Secondary objectives are the exploration of pharmacokinetics (PK) of BI 764198 after single and multiple oral dosing.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects according to the assessment of the investigator, as based on a complete medical history, including a physical examination, vital signs (BP, PR), 12-lead ECG, and clinical laboratory tests
* Japanese ethnicity, according to the following criteria: born in Japan, have lived outside of Japan <10 years, and have parents and grandparents who are Japanese
* Age of 20 to 45 years at screening (inclusive)
* BMI of 18.5 to 25.0 kg/m2 (inclusive)
* Signed and dated written informed consent prior to admission to the trial, in accordance with GCP and local legislation
* Willingness to comply with contraception requirements. Subjects who are sexually active must use adequate contraception methods throughout the trial and until three months after the last administration of trial medication. Adequate methods are:

  * A vasectomy performed at least 1 year prior to screening and with medical assessment of the surgical success or
  * Surgical sterilisation, including bilateral tubal occlusion, hysterectomy or bilateral oophorectomy, of the subject's female partner or
  * The use of condoms, if the female partner uses an adequate contraception method in addition, e.g., intrauterine device (IUD), or hormonal contraception, such as implants and injectables*, combined with oral or vaginal contraceptives, that started at least 2 months prior to first drug administration, or barrier method, e.g., diaphragm with spermicide* * hormonal contraception via implants and injectables, and diaphragm with spermicide are not approved in Japan Unprotected sexual intercourse with a pregnant partner is not allowed throughout the trial and until three months after the last administration of trial medication.

Exclusion Criteria:

* Any finding in the medical examination (including BP, PR or ECG) deviating from normal and assessed as clinically relevant by the investigator
* Repeated measurement of systolic blood pressure outside the range of 90 to 140 mmHg, diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 50 to 90 bpm
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Any evidence of a concomitant disease assessed as clinically relevant by the investigator
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Cholecystectomy or other surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy or simple hernia repair)- Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
* History of relevant orthostatic hypotension, fainting spells, or blackouts Further exclusion criteria apply.

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2021-02-06 (Actual); Primary Completion 2021-10-16 (Actual); Study Completion 2021-10-16 (Actual)

PRIMARY OUTCOMES:
The percentage [%] of subjects with drug-related adverse events | Up to 34 days

SECONDARY OUTCOMES:
After single dose: AUC0-∞ (area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity) | Up to 6 days
After single dose: Cmax (maximum measured concentration of the analyte in plasma) | Up to 6 days
After the last dose of multiple dose segment: AUCτ,ss (area under the concentration-time curve of the analyte in plasma at steady state over a uniform dosing interval τ) | Up to 22 days
After the last dose of multiple dose segment: Cmax,ss (maximum measured concentration of the analyte in plasma at steady state over a uniform dosing interval τ) | Up to 22 days

CONTACTS AND LOCATIONS:
Locations (1):
- SOUSEIKAI Sumida Hospital, Tokyo, Sumida-ku, Japan

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents, except for the following exclusions:
  1. studies in products where Boehringer Ingelheim is not the license holder;
  2. studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials;
  3. studies conducted in a single center or targeting rare diseases (because of limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- [Derived] Yonemura T, Sarashina A, Tachibana Y, Retlich S, Soleymanlou N. A randomized, Phase I study of the safety, tolerability, and pharmacokinetics of BI 764198, a transient receptor potential channel 6 (TRPC6) inhibitor, in healthy Japanese men. Expert Opin Investig Drugs. 2025 May;34(5):425-433. doi: 10.1080/13543784.2025.2510664. Epub 2025 Jun 3. PMID 40402558
- See also: Related Info — http://www.mystudywindow.com